CLINICAL TRIAL: NCT03588702
Title: Clinical Evaluation of the Safety and Performance of RF and PEMF Following Liposuction
Brief Title: RF and PEMF Following Liposuction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0817
Record Dates: First submitted 2018-07-03; First posted 2018-07-17 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Lipolysis
Keywords: radiofrequency; pulsed electro-magnetic fields; liposuction

STUDY DESIGN:
Intervention Model Description: Subjects act as their own control.
Masking Description: Independent blinded reviewers to view photographs to assess improvement of skin appearance of the treated side at 1 month post-treatment using the General Aesthetic Improvement Scale (GAIS) compared to the non-treated side
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venus Legacy LB2 Body applicator group (Experimental): Liposuction area is divided into 2 equal sections. One section receives RF and PEMF treatment.
  Interventions: Device: RF and PEMF treatment

INTERVENTIONS:
Device: RF and PEMF treatment — Treatment with Venus Legacy LB2 body applicator
  Other Names: Venus Legacy LB2 Body applicator

SUMMARY:
The Venus Legacy LB2 Body applicator is intended for circumference reduction treatment by reducing fat cell size and enhancing collagen synthesis as the result of thermal and non-thermal collagen stimulation. This is an open-label, evaluator-blind study of the safety and performance of radiofrequency (RF) and pulsed electromagnetic field (PEMF) therapy following liposuction. The study will enroll up to 50 male and female subjects requesting treatment of the back, flanks and/or thighs to improve appearance following liposuction. Subjects will receive a total of six study treatments to one side of their body (back, flanks and/or thighs) at one week intervals. Subjects will be followed up at one month after their last study treatment. Treatment outcomes will be compared to the non-treated side.

DETAILED DESCRIPTION:
Adipose tissue is a loose type of connective tissue specialized to store lipids. The majority of lipids stored in adipose cells are triglycerides formed from imported free fatty acids and glycerol. It is not uniformly distributed in the body. The major adipose depot is subcutaneous (about 80% of all body fat).

The technology options for skin tightening and body contouring have included vacuum massage, infrared laser energy, high frequency focused ultrasound, cryolipolysis, radiofrequency energy and various hybrid energy device options. Radiofrequency energy devices have remained the most common and dominant technology in the noninvasive management of skin tightening, cellulite improvement and body contouring enhancement, as they can treat all these conditions with relatively consistent results.

The RF energy is high frequency alternating electrical current that passes into the dermis and hypodermal tissues without disruption of the epidermal-dermal barrier. The high frequency oscillating electrical current results in collisions between charged molecules and ions and the micromolecular mechanical energy from these collisions is transformed into heat. This biological RF heat occurs irrespective of chromophore or skin type and is not dependent upon selective photothermolysis. The RF heat has different biological and hence, clinical effects, depending upon the tissue targeted. In the dermis, where the primary cellular element is the fibroblast and the extracellular matrix (ECM) is comprised of collagen, elastin and ground substances, the RF mediated thermal stimulation of the ECM results in an immediate and temporary shrinkage of the collagen triple helix. Further, the RF thermal stimulation results in a microinflammatory stimulation of the fibroblast which in response produces new collagen (neocollagenesis) and new elastin neoelastogenesis), and ground substances. RF thermal stimulation of adipose tissue results in a thermal mediated stimulation and augmented activity of lipase mediated enzymatic degradation of adipocyte derived triglycerides into free fatty acids and glycerol. This amplification of the physiologic breakdown and egress of the triglycerides out of the adipocyte, while keeping the adipocyte cell membrane and cell function intact, results in RF induced shrinkage of the fat cells and body contouring.

The Venus Legacy LB2 Body Applicator Combines Multi-Polar RF current and Pulsed Electromagnetic Fields (PEMF) in synergy with suction/vacuum. PEMF has been shown to increase fibroblast derived collagen production through a non-thermal mechanism of membrane stimulation, and the stimulation of fibroblast mediated angiogenesis which facilitates and enhances wound healing in tissues. Theoretically then, the synergistic RF and PEMF would create RF thermal collagen stimulation and PEMF non-thermal stimulation of collagen, RF thermally mediated reduction in adipocyte size and PEMF micro-tissue healing effects to minimize edema, swelling and downtime that are associated with pure RF thermal therapies.

The objective of this clinical study is to evaluate the safety and performance of RF and PEMF using the Venus Legacy LB2 body applicator following liposuction to the back, flanks and/or thighs.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female older than 18 years of age but not older than 65 years of age.
2. Having suitable area for treatment (bilateral liposuction of the back, flanks or thighs performed 8 weeks prior to study).
3. BMI score is greater than 18.5 and less than 29.9.
4. Willingness to refrain from a change in diet/drinking/exercise/medication regimen for the entire course of the study.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth (vaginal birth or Caesarean surgery) less than 9 months ago, and/or breastfeeding.
2. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
3. Having a permanent implant in the treated areas, such as metal plates and screws or an injected chemical substance.
4. Having undergone any other surgery in the treated areas within 9 months of treatment or during the study.
5. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
6. Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders.
7. Having a known anti-coagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course.
8. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
9. Suffering from hormonal imbalance which may affect weight or cellulite.
10. History of significant lymphatic drainage problems.
11. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment or during the treatment course.
12. History of keloid scarring or of abnormal wound healing.
13. History of being especially prone to bruising.
14. History of epidermal or dermal disorders (particularly if involving collagen or micro-vascularity).
15. Use of oral retinoids (e.g. isotretinoin (Accutane®)) within 6 months of treatment or during the study.
16. Use of anti-cellulite creams within a month of treatment or during the course of the study.
17. Significant change in diet or exercise regimen within a month of enrollment or during this study and/or weight loss or gain of 10 lbs. (4.5 kgs) within 2 months of enrollment or during this study.
18. Participation in a study of another device or drug within 1 month prior to enrollment or during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Improvement in skin appearance of the treated side | One month after last treatment
  Using the General Aesthetic improvement scale (GAIS), blinded reviewers assess photos of liposuction area to determine improvement in treated side as compared to non-treated side where 3 is very much improved; 2 is much improved; 1 is imporved; 0 is no change; -1 is worse; -2 is much worse and -3 is very much worse.

SECONDARY OUTCOMES:
Improvement in skin elasticity of the treated side | One month after last treatment
  As measured by a cutometer, determine improvement in skin elasticity of the treated side as compared to the non-treated side where parameter R2, gross elasticity is used. The closer the value is to 1 (100%), the more elastic the skin.
Subject satisfaction of treatment | One month after last treatment
  Using the 5-point Likert Satisfaction scale, subjects indicate their satisfaction with the appearance of the treated side as compared to non-treated side where 0 is very unsatisfied; 1 is unsatisfied; 2 is having no opinion; 3 is satisfied and 4 is very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cardarelli, Study Director — Venus Concept
Locations (1):
- Ocean Clinic, Marbella, Spain